CLINICAL TRIAL: NCT06886776
Title: Implementing a Secure Firearm Storage Program in Illinois Health Centers in Partnership with AllianceChicago and the Illinois Primary Health Care Association (COMMUNITY ASPIRE)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: AllianceChicago (Other); Illinois Primary Health Care Association (Unknown); University of Pennsylvania (Other); National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Rinad Beidas, Ralph Seal Paffenbarger Professor and Chair, Department of Medical Social Sciences, Northwestern University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: FP00003311; R01NR021291 (NIH)
Record Dates: First submitted 2025-03-14; First posted 2025-03-20 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Suicide
Keywords: Implementation science; Firearms; Suicide; Pediatrics; Federally qualified health centers
MeSH Terms: conditions — Suicide

STUDY DESIGN:
Intervention Model Description: Stepped wedge randomized controlled trial
Masking Description: Data analyst and biostatistician will be blinded to randomization assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Baseline/usual care (No Intervention): During the baseline data collection phase, no individuals will be exposed to S.A.F.E. Firearm. No training or facilitation will be received. The length of the baseline data collection phase will differ between each "wedge" (i.e., group of clinics) depending on when the group is randomly assigned to cross over into the implementation phase. All sites will be in the baseline data collection phase for at least six months before having the interventions activated.
- Implementation phase (training and facilitation received, S.A.F.E. Firearm delivered) (Experimental): Once a group of clinics crosses over from the baseline data collection phase, the implementation approaches (e.g., training, facilitation) and the S.A.F.E. Firearm program will be enacted. S.A.F.E. Firearm involves pediatric clinicians having a secure firearm storage discussion with a parent or guardian during their child's well-visit and offering them a free cable firearm lock. This implementation phase will last for 12 months.
  Interventions: Behavioral: Implementation package (training and facilitation)
- Sustainment (training and facilitation removed) (No Intervention): Following the conclusion of the 12 months in which the implementation approaches (training and facilitation) are used at a clinic, outcomes will be assessed for the duration of the study during a "sustainment" window.
  No additional training or facilitation will be received during the sustainment period following the experimental period. However, clinics will still continue to deliver S.A.F.E. Firearm.

INTERVENTIONS:
Behavioral: Implementation package (training and facilitation) — Training includes an initial presentation on S.A.F.E. Firearm, S.A.F.E. Firearm informational guides and other resources to support delivery, and recommendations for additional, optional self-guided learning resources.
  Facilitation will last twelve months at each site. It may involve 1) a pre-implementation readiness assessment for each clinic to identify potential implementation barriers and develop relationships with constituents; 2) kick-off meetings at the launch of the trial, at which clinic staff will identify how and where S.A.F.E. Firearm will be implemented within the clinic; 3) goal-setting within the first few months of the program; 4) trouble-shooting to address barriers identified during the pre-implementation readiness assessment and emergent challenges; and 5) designing a sustainment plan to maintain S.A.F.E. Firearm for future years.
  Arms: Implementation phase (training and facilitation received, S.A.F.E. Firearm delivered)

SUMMARY:
This randomized controlled trial will take place in up to 15 community health centers across the state of Illinois. Researchers will be studying S.A.F.E. Firearm, a program that aims to increase secure storage of firearms in homes with children. Specifically, S.A.F.E. Firearm includes a brief conversation between pediatric clinicians and parents about secure firearm storage and an offer of a free cable firearm lock within the well-child visit. Researchers will also study a package of strategies to help pediatric clinics incorporate this new practice. The strategies include training for clinic personnel and facilitation, or tailored problem-solving support.

The questions the study aims to answer are:

* How effective is the package of strategies at helping pediatric clinics adopt this new practice?
* How effective is the S.A.F.E. Firearm program at changing parents' and guardians' firearm storage behavior?

Some parents and guardians will be invited to complete a brief survey after their visit about their experiences receiving S.A.F.E. Firearm. Some community health center personnel will also be invited to complete an interview about their experiences with S.A.F.E. Firearm and the package of strategies.

DETAILED DESCRIPTION:
While some large health systems have successfully adopted secure firearm storage programs such as S.A.F.E. Firearm into routine practice, there is limited research on the implementation of secure firearm storage programs in community settings, such as community health centers, which serve large populations of Americans. These settings often face challenges such as financial pressures and high staff turnover, which were made worse by the COVID-19 pandemic. Therefore, before deploying a secure firearm storage program in this new setting, adaptation is needed. As part of Aim 1 of the grant funding this project, the research team is working with local community-based organizations, firearm safety experts, community health center personnel, and parents and guardians (hereafter, "parents") to understand the changes that need to be made to the S.A.F.E. Firearm program and the package of implementation strategies that have been successfully used in previous studies to help pediatric clinics adopt this new practice (training, facilitation, other strategies selected in tandem with partners in the adaptation process). The research team will incorporate needed changes before the present trial will begin.

In the present study, the research team will conduct a hybrid type III effectiveness-implementation trial to test the effect of the adapted S.A.F.E. Firearm program and associated strategies. The trial will be conducted across pediatric well-visits in community health centers across the state of Illinois using a stepped wedge design. Clinics will be randomized into clusters of clinics and the implementation approach (staff training, facilitation, other strategies selected in tandem with partners in the adaptation process) will be activated upon the start of each step.

Aims for the study include:

Aim 2. We will conduct a pragmatic hybrid type III stepped wedge effectiveness-implementation randomized controlled trial with community health centers across Illinois to test the effectiveness of our adapted implementation approach (training and facilitation emphasizing S.A.F.E. Firearm delivery) on parent-reported receipt of S.A.F.E. Firearm (i.e., reach; primary implementation outcome). We will also assess secondary implementation outcomes (stage of implementation, cost, acceptability) and effectiveness outcomes (parent firearm storage behavior).

Aim 3. We will use mixed methods to identify mechanisms. First, we will conduct interviews to understand constituent perspectives on implementation mechanisms and equitable intervention receipt. Second, we will evaluate reach and firearm storage behavior by demographic characteristics and social determinants of health.

ELIGIBILITY:
Inclusion Criteria:

Parent participants

* Be a parent of a child ages 0-17 who has a well-visit at a participating health care clinic in the state of Illinois
* Attend the child's well-visit

Health care personnel

* Be employed at a participating health care clinic in the state of Illinois
* Aged 18+ years

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 666 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2028-08-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Parent-reported reach of S.A.F.E. Firearm | Reach will be collected via survey sent to parents after well-visits for the 3-year study period (baseline through sustainment phases)
  The proportion of eligible pediatric well-visits for which parents report receiving the two components of S.A.F.E. Firearm (discussion of secure firearm storage, offer of a free cable firearm lock)

CONTACTS AND LOCATIONS:
Locations (1):
- Illinois Primary Health Care Association, Springfield, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided